CLINICAL TRIAL: NCT01248949
Title: Phase 1/1b, Open-Label, Dose-Escalation and Expansion Study to Evaluate the Safety and Antitumor Activity of MEDI3617 as a Single-Agent or in Combination Therapy in Adult Subjects With Advanced Solid Tumors
Brief Title: A Study to Evaluate the Safety and Antitumor Activity in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD-ON-MEDI3617-1043
Record Dates: First submitted 2010-11-23; First posted 2010-11-25 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Advanced Solid Tumors; Advanced Recurrent Ovarian Tumors
Keywords: Advanced solid tumors; Advanced recurrent ovarian tumors; MEDI3617; Ang2; Ovarian cancer; Malignant glioma
MeSH Terms: conditions — Ovarian Neoplasms; Glioma | interventions — MEDI3617; Bevacizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- MEDI3617 SINGLE AGENT TOTAL (Experimental): Participants will receive MEDI3617 via intravenous (IV) infusion every 3 weeks (Q3W) in each cycle until unacceptable toxicity, initiation of alternative anticancer treatment, documented disease progression, or other reasons. Each cycle consists of 21 days.
  Interventions: Drug: MEDI3617
- MEDI3617 + BEVACIZUMAB Q3W ESCALATION (Experimental): Participants will receive MEDI3617 with bevacizumab via IV infusion every 3 weeks (Q3W) in each cycle until unacceptable toxicity, initiation of alternative anticancer treatment, documented disease progression, or other reasons. Each cycle consists of 21 days.
  Interventions: Drug: MEDI3617; Drug: Bevacizumab
- MEDI3617 + BEVACIZUMAB Q2W TOTAL (Experimental): Participants will receive MEDI3617 with bevacizumab via IV infusion every 2 weeks (Q2W) in each cycle until unacceptable toxicity, initiation of alternative anticancer treatment, documented disease progression, or other reasons. Each cycle consists of 28 days.
  Interventions: Drug: MEDI3617; Drug: Bevacizumab
- MEDI3617 + PACLITAXEL TOTAL (Experimental): Participants will receive MEDI3617 on Days 1 and 15 with paclitaxel on Days 1, 8, and 15 via IV infusion in each cycle until unacceptable toxicity, documented disease progression, or other reasons. Each cycle consists of 28 days.
  Interventions: Drug: MEDI3617; Drug: Paclitaxel
- MEDI3617 + CARBOPLATIN/PACLITAXEL TOTAL (Experimental): Participants will receive MEDI3617 with carboplatin and paclitaxel on Day 1 via IV infusion in each cycle until unacceptable toxicity, documentation of disease progression, or other reasons. Each cycle consists of 21 days.
  Interventions: Drug: MEDI3617; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: MEDI3617 — Participants will receive MEDI3617 via IV infusion in each cycle until unacceptable toxicity, initiation of alternative anticancer treatment, documented disease progression, or other reasons.
Drug: Bevacizumab — Participants will receive bevacizumab via IV infusion in each cycle until unacceptable toxicity, initiation of alternative anticancer treatment, documented disease progression, or other reasons.
  Arms: MEDI3617 + BEVACIZUMAB Q2W TOTAL; MEDI3617 + BEVACIZUMAB Q3W ESCALATION
Drug: Paclitaxel — Participants will receive paclitaxel via IV infusion in each cycle until unacceptable toxicity, documented disease progression, or other reasons.
  Arms: MEDI3617 + CARBOPLATIN/PACLITAXEL TOTAL; MEDI3617 + PACLITAXEL TOTAL
Drug: Carboplatin — Participants will receive carboplatin via IV infusion in each cycle until unacceptable toxicity, documentation of disease progression, or other reasons.
  Arms: MEDI3617 + CARBOPLATIN/PACLITAXEL TOTAL

SUMMARY:
To determine the maximum tolerated dose or optimal biological dose, and the safety profile of MEDI3617 when given as a single-agent or in combination with other chemotherapeutic agents in subjects with advanced solid malignancies resistant to standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of advanced solid tumors (dose-escalation phase) or another solid tumor type based on antitumoral activity (dose-expansion phase) that are not responsive to standard therapy or for which no standard therapy exists
* Patients must be 18 years of age or older
* Karnofsky Performance Status ≥ 70
* Toxicities from previous cancer therapies must have recovered to CTCAE Grade = or < 2
* Adequate organ and marrow function
* Using adequate contraceptive measures, be surgically sterile or post-menopausal

Exclusion Criteria:

* Concurrently enrolled in another clinical study, except for non-interventiona observational studies, or if in a follow up period from a previous study
* Receipt of any investigational anticancer therapy within 30 days prior to the first dose of MEDI3617, or in the case of monoclonal antibodies (eg, bevacizumab), 42 days prior to the first dose of MEDI3617
* Current or previous treatment with angiopoietin inhibitors, or inhibitors of Tie1 or Tie2 including, but not limited to, AMG386, CVX-060, XL880, and XL820
* Any concurrent chemotherapy, radiotherapy, immunotherapy, biologic or hormonal therapy for cancer treatment
* Use of immunosuppressive medication or systemic steroids within 7 days prior to first dose of MEDI3617
* Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results
* Known bleeding diathesis
* Pulmonary hemorrhage or gross hemoptysis within 6 months prior to enrollment
* Therapeutic or palliative radiation therapy within 2 weeks prior to enrollment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2010-10; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune, LLC, Study Director — MedImmune LLC
Locations (10):
- United States (10):
  - Research Site, Los Angeles, California
  - Research Site, Stanford, California
  - Research Site, Lafayette, Indiana
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Buffalo, New York
  - Research Site, New York, New York
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 162 participants were screened, of which 46 did not meet eligibility criteria and were considered as screen failures; the remaining 116 participants entered into the study and treated with MEDI3617.
Groups:
- MEDI3617 SINGLE AGENT TOTAL: Participants received MEDI3617 via IV infusion every 3 weeks (Q3W) in each cycle until unacceptable toxicity, initiation of alternative anticancer treatment, documented disease progression, or other reasons. Each cycle consists of 21 days.
- MEDI3617 + BEVACIZUMAB Q3W ESCALATION TOTAL: Participants received MEDI3617 with bevacizumab via IV infusion every 3 weeks (Q3W) in each cycle until unacceptable toxicity, initiation of alternative anticancer treatment, documented disease progression, or other reasons. Each cycle consists of 21 days.
- MEDI3617 + BEVACIZUMAB Q2W TOTAL: Participants received MEDI3617 with bevacizumab via IV infusion every 2 weeks (Q2W) in each cycle until unacceptable toxicity, initiation of alternative anticancer treatment, documented disease progression, or other reasons. Each cycle consists of 28 days.
- MEDI3617 + PACLITAXEL TOTAL: Participants received MEDI3617 on Days 1 and 15 with paclitaxel on Days 1, 8, and 15 via IV infusion in each cycle until unacceptable toxicity, documented disease progression, or other reasons. Each cycle consists of 28 days.
- MEDI3617 + CARBOPLATIN/ PACLITAXEL TOTAL: Participants received MEDI3617 with carboplatin and paclitaxel on Day 1 via IV infusion in each cycle until unacceptable toxicity, documentation of disease progression, or other reasons. Each cycle consists of 21 days.
Period: Overall Study
Arm/Group | MEDI3617 SINGLE AGENT TOTAL | MEDI3617 + BEVACIZUMAB Q3W ESCALATION TOTAL | MEDI3617 + BEVACIZUMAB Q2W TOTAL | MEDI3617 + PACLITAXEL TOTAL | MEDI3617 + CARBOPLATIN/ PACLITAXEL TOTAL
Started | 42 | 16 | 38 | 13 | 7
Completed | 9 | 3 | 1 | 3 | 3
Not Completed | 33 | 13 | 37 | 10 | 4
Not completed — Lost to Follow-up | 2 | 2 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 5 | 3 | 11 | 3 | 1
Not completed — Death | 22 | 7 | 21 | 6 | 2
Not completed — Alternative Therapy | 1 | 0 | 0 | 0 | 0
Not completed — Alternative Therapy. | 1 | 0 | 0 | 0 | 0
Not completed — Palliative Radiation To Brain Metastases | 1 | 0 | 0 | 0 | 0
Not completed — Entered Hospice And Refused Follow Up | 0 | 0 | 0 | 0 | 1
Not completed — Participant Went To Hospice | 0 | 0 | 1 | 0 | 0
Not completed — Per Sponsor Request o Discontinue Drug | 1 | 0 | 0 | 0 | 0
Not completed — Pi Decision Due To Declining Status | 0 | 0 | 1 | 0 | 0
Not completed — Pi Discretion Due To Hospitalisation | 0 | 1 | 0 | 0 | 0
Not completed — Lesion In ThoracicSpine Requires Therapy | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who receive any treatment with MEDI3617.
Groups:
- MEDI3617 + CARBOPLATIN/PACLITAXEL TOTAL: Participants received MEDI3617 with carboplatin and paclitaxel on Day 1 via IV infusion in each cycle until unacceptable toxicity, documentation of disease progression, or other reasons. Each cycle consists of 21 days.
- Total: Total of all reporting groups
Arm/Group | MEDI3617 SINGLE AGENT TOTAL | MEDI3617 + BEVACIZUMAB Q3W ESCALATION TOTAL | MEDI3617 + BEVACIZUMAB Q2W TOTAL | MEDI3617 + PACLITAXEL TOTAL | MEDI3617 + CARBOPLATIN/PACLITAXEL TOTAL | Total
Number analyzed (Participants) | 42 | 16 | 38 | 13 | 7 | 116
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.4 (12.4) | 57.4 (11.9) | 57.7 (11.2) | 60.4 (12.7) | 56.7 (12.3) | 59.2 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 7 | 18 | 8 | 5 | 65
  Male | 15 | 9 | 20 | 5 | 2 | 51

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT was defined as any treatment-related, grade 3 or higher toxicity (according to the National Cancer Institute's Common Terminology Criteria for Adverse Events [NCI CTCAE] version 4.0); occurring during the first 21 or 28 days after the initial administration of MEDI3617.
Time Frame: From the time of first administration of MEDI3617 single agent or MEDI3617 combination therapy through the first 21-day or 28-day cycle (Cycle 1)
Population: DLT Evaluable population included all participants enrolled in dose-escalation, who received at least 1 full assigned dose of single-agent MEDI3617 or full assigned doses of MEDI3617 and standard therapeutic agents on Cycle 1 and completed safety follow-up or experienced a DLT at any point during the 21-day or 28-day DLT evaluation period.
Measure: Number; unit: Participants
Arm/Group | MEDI3617 SINGLE AGENT TOTAL | MEDI3617 + BEVACIZUMAB Q3W ESCALATION TOTAL | MEDI3617 + BEVACIZUMAB Q2W TOTAL | MEDI3617 + PACLITAXEL TOTAL | MEDI3617 + CARBOPLATIN/PACLITAXEL TOTAL
Number analyzed (Participants) | 23 | 15 | 22 | 11 | 6
Participants | 1 | 1 | 2 | 1 | 1

2. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The dose-escalation phase used a 3 + 3 design. If greater than or equal to 2 (≥ 2) participants in a dose cohort experienced a DLT during the DLT period, the MTD was exceeded and no further participants were enrolled into that dose cohort. If this occurred, the preceding dose cohort was evaluated for the MTD and a total of 6 participants were treated at the preceding dose. If less than or equal to 1 (≤ 1) of 6 participants experienced a DLT at the preceding dose, then this dose level was the MTD. DLTs were defined as any treatment-related, grade 3 or higher toxicity (according to the National Cancer Institute's Common Terminology Criteria for Adverse Events [NCI CTCAE] version 4.0); occurring during the first 21 or 28 days after the initial administration of MEDI3617.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: milligram (mg)
Arm/Group | MEDI3617 SINGLE AGENT TOTAL | MEDI3617 + BEVACIZUMAB Q3W ESCALATION TOTAL | MEDI3617 + BEVACIZUMAB Q2W TOTAL | MEDI3617 + PACLITAXEL TOTAL | MEDI3617 + CARBOPLATIN/PACLITAXEL TOTAL
Number analyzed (Participants) | 23 | 15 | 22 | 11 | 6
milligram (mg) | NA — The highest dose level was cleared and the MTD was not reached. | NA — A DLT was reported at the highest dose level, but only 5 out of the 6 participants enrolled were evaluable for DLT. Thus, it is unclear if the MTD was exceeded or reached at the highest dose level tested. | NA — The highest dose level was cleared and the MTD was not reached. | NA — The highest dose level was cleared and the MTD was not reached. | NA — A DLT was reported at the highest dose level, but it is unclear if the MTD was exceeded or reached, as only 3 participants were enrolled (all participants were evaluable for DLT).

3. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant administered investigational product and which does not necessarily have a causal relationship with this treatment. A serious adverse event (SAE) was an AE resulting in any of following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs were events occurring after administration of investigational product.
Time Frame: From start of study drug administration up to 90 days after the last dose of MEDI3617
Population: Safety population included all participants who received treatment with MEDI3617.
Measure: Number; unit: Participants
Arm/Group | MEDI3617 SINGLE AGENT TOTAL | MEDI3617 + BEVACIZUMAB Q3W ESCALATION TOTAL | MEDI3617 + BEVACIZUMAB Q2W TOTAL | MEDI3617 + PACLITAXEL TOTAL | MEDI3617 + CARBOPLATIN/PACLITAXEL TOTAL
Number analyzed (Participants) | 42 | 16 | 38 | 13 | 7
Participants
  TEAEs | 42 | 16 | 38 | 13 | 7
  TESAEs | 18 | 4 | 18 | 7 | 4

4. Primary Outcome: Number of Participants With Laboratory Abnormalities Recorded as Adverse Events (AEs)
Description: Laboratory evaluations were performed, including hematology and serum chemistry. An AE was any untoward medical occurrence in a participant administered investigational product and which does not necessarily have a causal relationship with this treatment. AEs related to laboratory abnormalities were recorded and reported.
Time Frame: From start of study drug administration up to 90 days after the last dose of MEDI3617
Population: Safety population included all participants who received treatment with MEDI3617.
Measure: Number; unit: Participants
Arm/Group | MEDI3617 SINGLE AGENT TOTAL | MEDI3617 + BEVACIZUMAB Q3W ESCALATION TOTAL | MEDI3617 + BEVACIZUMAB Q2W TOTAL | MEDI3617 + PACLITAXEL TOTAL | MEDI3617 + CARBOPLATIN/PACLITAXEL TOTAL
Number analyzed (Participants) | 42 | 16 | 38 | 13 | 7
Participants
  Hematology: Anemia | 5 | 1 | 1 | 3 | 2
  Hematology: Leukopenia | 0 | 0 | 0 | 1 | 2
  Hematology: Neutropenia | 1 | 0 | 0 | 0 | 3
  Hematology: Thombocytopenia | 0 | 0 | 0 | 0 | 2
  Hematology: White blood cell count decreased | 2 | 0 | 0 | 0 | 1
  SerChem: Alanine aminotransferase increased | 0 | 0 | 1 | 0 | 0
  SerChem: Aspartate aminotransferase increased | 0 | 1 | 2 | 1 | 0
  SerChem: Blood alkaline phosphatase increased | 1 | 0 | 1 | 1 | 0
  SerChem: Blood creatinine increased | 2 | 1 | 2 | 1 | 0
  SerChem: Blood lactate dehydrogenase increased | 0 | 0 | 0 | 1 | 0
  SerChem: Blood potassium increased | 0 | 1 | 0 | 0 | 0
  SerChem: Blood triglycerides increased | 0 | 1 | 1 | 0 | 0
  SerChem: Blood urea increased | 0 | 0 | 1 | 0 | 0
  SerChem: Gamma-glutamyltransferase increased | 1 | 1 | 1 | 1 | 0
  SerChem: Hyperglycaemia | 1 | 0 | 0 | 1 | 0
  SerChem: Hyperkalaemia | 1 | 0 | 0 | 0 | 0
  SerChem: Hypertriglyceridaemia | 0 | 1 | 0 | 0 | 0
  SerChem: Hyperuricaemia | 1 | 1 | 0 | 1 | 0
  SerChem: Hypoalbuminaemia | 0 | 1 | 1 | 0 | 0
  SerChem: Hypocalcaemia | 0 | 1 | 0 | 0 | 0
  SerChem: Hypoglycaemia | 1 | 1 | 2 | 0 | 0
  SerChem: Hypokalaemia | 3 | 0 | 2 | 0 | 1
  SerChem: Hypomagnesaemia | 1 | 1 | 0 | 1 | 3
  SerChem: Hyponatremia | 0 | 2 | 1 | 1 | 2

5. Primary Outcome: Number of Participants With Vital Sign Abnormalities Recorded as Adverse Events (AEs)
Description: Vital signs included parameters such as heart rate, blood pressure, temperature, weight and respiratory rate. An AE was any untoward medical occurrence in a participant administered investigational product and which does not necessarily have a causal relationship with this treatment. AEs related to vital signs abnormalities were recorded and reported.
Time Frame: From start of study drug administration up to 90 days after the last dose of MEDI3617
Population: Safety population included all participants who received treatment with MEDI3617.
Measure: Number; unit: Participants
Arm/Group | MEDI3617 SINGLE AGENT TOTAL | MEDI3617 + BEVACIZUMAB Q3W ESCALATION TOTAL | MEDI3617 + BEVACIZUMAB Q2W TOTAL | MEDI3617 + PACLITAXEL TOTAL | MEDI3617 + CARBOPLATIN/PACLITAXEL TOTAL
Number analyzed (Participants) | 42 | 16 | 38 | 13 | 7
Participants
  Arrhythmia | 1 | 0 | 0 | 0 | 0
  Sinus tachycardia | 0 | 1 | 0 | 1 | 0
  Tachycardia | 1 | 1 | 0 | 1 | 0
  Pyrexia | 3 | 3 | 1 | 0 | 1
  Weight decreased | 0 | 2 | 0 | 0 | 1
  Weight increased | 9 | 2 | 0 | 1 | 0
  Hypertension | 10 | 7 | 13 | 3 | 2
  Hypotension | 0 | 0 | 1 | 0 | 0

6. Primary Outcome: Number of Participants With Echocardiogram Abnormalities Recorded as Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant administered investigational product and which does not necessarily have a causal relationship with this treatment. AEs related to echocardiogram abnormalities were recorded and reported. The only AE reported was ejection fraction decreased in the MEDI3617 + Paclitaxel total group.
Time Frame: From start of study drug administration up to 90 days after the last dose of MEDI3617
Population: Safety population included all participants who received treatment with MEDI3617.
Measure: Number; unit: Participants
Arm/Group | MEDI3617 SINGLE AGENT TOTAL | MEDI3617 + BEVACIZUMAB Q3W ESCALATION TOTAL | MEDI3617 + BEVACIZUMAB Q2W TOTAL | MEDI3617 + PACLITAXEL TOTAL | MEDI3617 + CARBOPLATIN/PACLITAXEL TOTAL
Number analyzed (Participants) | 42 | 16 | 38 | 13 | 7
Participants | 0 | 0 | 0 | 1 | 0

7. Primary Outcome: Number of Participants With Electrocardiogram Abnormalities Recorded as Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant administered investigational product and which does not necessarily have a causal relationship with this treatment. AEs related to electrocardiogram abnormalities were recorded and reported. The only AE reported was electrocardiogram QT prolonged in the MEDI3617 + Bevacizumab Q2W total group.
Time Frame: From start of study drug administration up to 90 days after the last dose of MEDI3617
Population: Safety population included all participants who received treatment with MEDI3617
Measure: Number; unit: Participants
Arm/Group | MEDI3617 SINGLE AGENT TOTAL | MEDI3617 + BEVACIZUMAB Q3W ESCALATION TOTAL | MEDI3617 + BEVACIZUMAB Q2W TOTAL | MEDI3617 + PACLITAXEL TOTAL | MEDI3617 + CARBOPLATIN/PACLITAXEL TOTAL
Number analyzed (Participants) | 42 | 16 | 38 | 13 | 7
Participants | 0 | 0 | 1 | 0 | 0

8. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of MEDI3617
Description: Cmax is the maximum observed serum concentration of MEDI3617. Here, "n" is number of participants analyzed for this endpoint at a specific dose.
Time Frame: Days 1, 2 (MEDI3617 single agent only), 4, 8, 15 (Cycle 1); Day 1 (Cycle 2 and every cycle after), Day 15 (MEDI3617 + bev Q2W and MEDI3617 + paclitaxel only, Cycle 2 and every cycle after); end of treatment; 30 days and 3 months post last dose
Population: All participants who received treatment with MEDI3617 and for whom PK blood samples were collected and evaluated.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/ml)
Arm/Group | MEDI3617 SINGLE AGENT TOTAL | MEDI3617 + BEVACIZUMAB Q3W ESCALATION TOTAL | MEDI3617 + BEVACIZUMAB Q2W TOTAL | MEDI3617 + PACLITAXEL TOTAL | MEDI3617 + CARBOPLATIN/PACLITAXEL TOTAL
Number analyzed (Participants) | 41 | 16 | 35 | 13 | 7
microgram per milliliter (mcg/ml)
  Cohort -2 (n=3) | 1.39 (0.254) | NA (NA) — Cohort -2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort -2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort -2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort -2 was part of the MEDI3617 Single agent total group.
  Cohort -1 (n=2) | 2.44 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort -1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort -1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort -1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort -1 was part of the MEDI3617 Single agent total group.
  Cohort 1 (n=6) | 6.63 (3.48) | NA (NA) — Cohort 1 was part of the MEDI3617 Single agent total group | NA (NA) — Cohort 1 was part of the MEDI3617 Single agent total group | NA (NA) — Cohort 1 was part of the MEDI3617 Single agent total group | NA (NA) — Cohort 1 was part of the MEDI3617 Single agent total group
  Cohort 2 (n=3) | 50.2 (28.8) | NA (NA) — Cohort 2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 2 was part of the MEDI3617 Single agent total group.
  Cohort 3 (n=3) | 82.4 (2.68) | NA (NA) — Cohort 3 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 3 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 3 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 3 was part of the MEDI3617 Single agent total group.
  Cohort 4 (n=3) | 239 (79.5) | NA (NA) — Cohort 4 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 4 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 4 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 4 was part of the MEDI3617 Single agent total group.
  Cohort 5 (n=4) | 785 (189) | NA (NA) — Cohort 5 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 5 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 5 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 5 was part of the MEDI3617 Single agent total group.
  Cohort ovarian cancer expansion (OCE) -1 (n=15) | 336 (62.2) | NA (NA) — Cohort OCE -1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE -1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE -1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE -1 was part of the MEDI3617 Single agent total group.
  Cohort OCE 1 (n=2) | 346 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort OCE 1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE 1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE 1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE 1 was part of the MEDI3617 Single agent total group.
  Cohort MB 1A (n=4) | NA (NA) — Cohort MB 1A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | 30.4 (26.8) | NA (NA) — Cohort MB 1A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 1A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 1A was part of the MEDI3617 + Bevacizumab Q3W escalation group.
  Cohort MB 2A (n=3) | NA (NA) — Cohort MB 2A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | 55.3 (12.6) | NA (NA) — Cohort MB 2A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 2A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 2A was part of the MEDI3617 + Bevacizumab Q3W escalation group.
  Cohort MB 3A (n=3) | NA (NA) — Cohort MB 3A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | 235 (90.5) | NA (NA) — Cohort MB 3A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 3A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 3A was part of the MEDI3617 + Bevacizumab Q3W escalation group.
  Cohort MB 4A (n=6) | NA (NA) — Cohort MB 4A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | 348 (54.6) | NA (NA) — Cohort MB 4A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 4A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 4A was part of the MEDI3617 + Bevacizumab Q3W escalation group.
  Cohort MB 1B (n=7) | NA (NA) — Cohort MB 1B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 1B was part of the MEDI3617 + Bevacizumab Q2W Total group. | 44.5 (39.3) | NA (NA) — Cohort MB 1B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 1B was part of the MEDI3617 + Bevacizumab Q2W Total group.
  Cohort MB 2B (n=3) | NA (NA) — Cohort MB 2B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 2B was part of the MEDI3617 + Bevacizumab Q2W Total group. | 47.5 (23.3) | NA (NA) — Cohort MB 2B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 2B was part of the MEDI3617 + Bevacizumab Q2W Total group.
  Cohort MB 3B (n=8) | NA (NA) — Cohort MB 3B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 3B was part of the MEDI3617 + Bevacizumab Q2W Total group. | 116 (35.1) | NA (NA) — Cohort MB 3B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 3B was part of the MEDI3617 + Bevacizumab Q2W Total group.
  Cohort MB 4B (n=8) | NA (NA) — Cohort MB 4B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 4B was part of the MEDI3617 + Bevacizumab Q2W Total group. | 275 (86.2) | NA (NA) — Cohort MB 4B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 4B was part of the MEDI3617 + Bevacizumab Q2W Total group.
  Cohort TT2A (n=9) | NA (NA) — Cohort TT2A (participants with bevacizumab-refractory glioma), was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort TT2A (participants with bevacizumab-refractory glioma), was part of the MEDI3617 + Bevacizumab Q2W Total group. | 320 (170) | NA (NA) — Cohort TT2A (participants with bevacizumab-refractory glioma), was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort TT2A (participants with bevacizumab-refractory glioma), was part of the MEDI3617 + Bevacizumab Q2W Total group.
  Cohort MP1 (n=7) | NA (NA) — Cohort MP1 was part of the MEDI3617 + Paclitaxel group. | NA (NA) — Cohort MP1 was part of the MEDI3617 + Paclitaxel group. | NA (NA) — Cohort MP1 was part of the MEDI3617 + Paclitaxel group. | 114 (22.5) | NA (NA) — Cohort MP1 was part of the MEDI3617 + Paclitaxel group.
  Cohort MP2 (n=6) | NA (NA) — Cohort MP2 was part of the MEDI3617 + Paclitaxel group. | NA (NA) — Cohort MP2 was part of the MEDI3617 + Paclitaxel group. | NA (NA) — Cohort MP2 was part of the MEDI3617 + Paclitaxel group. | 209 (57.4) | NA (NA) — Cohort MP2 was part of the MEDI3617 + Paclitaxel group.
  Cohort MCP1 (n=4) | NA (NA) — Cohort MCP1 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP1 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP1 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP1 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | 200 (25.8)
  Cohort MCP2 (n=3) | NA (NA) — Cohort MCP2 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP2 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP2 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP2 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | 585 (491)

9. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC0-last) of MEDI3617
Description: AUC0-last is the Area Under the Concentration-Time Curve From Time Zero to the Time of the Last Quantifiable Concentration of MEDI3617. Here, "n" is number of participants analyzed for this endpoint at a specific dose.
Time Frame: as for outcome 8
Population: All participants who received treatment with MEDI3617 and for whom PK blood samples were collected and evaluated.
Measure: Mean (Standard Deviation); unit: day*mcg/mL
Arm/Group | MEDI3617 SINGLE AGENT TOTAL | MEDI3617 + BEVACIZUMAB Q3W ESCALATION TOTAL | MEDI3617 + BEVACIZUMAB Q2W TOTAL | MEDI3617 + PACLITAXEL TOTAL | MEDI3617 + CARBOPLATIN/PACLITAXEL TOTAL
Number analyzed (Participants) | 41 | 16 | 35 | 13 | 7
day*mcg/mL
  Cohort -2 (n=3) | 1.3 (0.429) | NA (NA) — Cohort -2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort -2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort -2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort -2 was part of the MEDI3617 Single agent total group.
  Cohort -1 (n=2) | 2.2 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort -1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort -1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort -1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort -1 was part of the MEDI3617 Single agent total group.
  Cohort 1 (n=6) | 11.9 (11.8) | NA (NA) — Cohort 1 was part of the MEDI3617 Single agent total group | NA (NA) — Cohort 1 was part of the MEDI3617 Single agent total group | NA (NA) — Cohort 1 was part of the MEDI3617 Single agent total group | NA (NA) — Cohort 1 was part of the MEDI3617 Single agent total group
  Cohort 2 (n=3) | 171 (69) | NA (NA) — Cohort 2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 2 was part of the MEDI3617 Single agent total group.
  Cohort 3 (n=3) | 438 (204) | NA (NA) — Cohort 3 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 3 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 3 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 3 was part of the MEDI3617 Single agent total group.
  Cohort 4 (n=3) | 2610 (1570) | NA (NA) — Cohort 4 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 4 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 4 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 4 was part of the MEDI3617 Single agent total group.
  Cohort 5 (n=4) | 3650 (2600) | NA (NA) — Cohort 5 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 5 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 5 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 5 was part of the MEDI3617 Single agent total group.
  Cohort OCE -1 (n=15) | 2610 (891) | NA (NA) — Cohort OCE -1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE -1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE -1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE -1 was part of the MEDI3617 Single agent total group.
  Cohort OCE 1 (n=2) | 2160 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort OCE 1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE 1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE 1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE 1 was part of the MEDI3617 Single agent total group.
  Cohort MB 1A (n=4) | NA (NA) — Cohort MB 1A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | 101 (48.8) | NA (NA) — Cohort MB 1A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 1A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 1A was part of the MEDI3617 + Bevacizumab Q3W escalation group.
  Cohort MB 2A (n=3) | NA (NA) — Cohort MB 2A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | 473 (223) | NA (NA) — Cohort MB 2A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 2A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 2A was part of the MEDI3617 + Bevacizumab Q3W escalation group.
  Cohort MB 3A (n=3) | NA (NA) — Cohort MB 3A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | 2280 (529) | NA (NA) — Cohort MB 3A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 3A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 3A was part of the MEDI3617 + Bevacizumab Q3W escalation group.
  Cohort MB 4A (n=6) | NA (NA) — Cohort MB 4A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | 2710 (1070) | NA (NA) — Cohort MB 4A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 4A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 4A was part of the MEDI3617 + Bevacizumab Q3W escalation group.
  Cohort MB 1B (n=7) | NA (NA) — Cohort MB 1B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 1B was part of the MEDI3617 + Bevacizumab Q2W Total group. | 94.7 (48.7) | NA (NA) — Cohort MB 1B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 1B was part of the MEDI3617 + Bevacizumab Q2W Total group.
  Cohort MB 2B (n=3) | NA (NA) — Cohort MB 2B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 2B was part of the MEDI3617 + Bevacizumab Q2W Total group. | 216 (61.8) | NA (NA) — Cohort MB 2B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 2B was part of the MEDI3617 + Bevacizumab Q2W Total group.
  Cohort MB 3B (n=8) | NA (NA) — Cohort MB 3B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 3B was part of the MEDI3617 + Bevacizumab Q2W Total group. | 805 (292) | NA (NA) — Cohort MB 3B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 3B was part of the MEDI3617 + Bevacizumab Q2W Total group.
  Cohort MB 4B (n=8) | NA (NA) — Cohort MB 4B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 4B was part of the MEDI3617 + Bevacizumab Q2W Total group. | 2310 (941) | NA (NA) — Cohort MB 4B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 4B was part of the MEDI3617 + Bevacizumab Q2W Total group.
  Cohort TT2A (n=9) | NA (NA) — Cohort TT2A (participants with bevacizumab-refractory glioma), was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort TT2A (participants with bevacizumab-refractory glioma), was part of the MEDI3617 + Bevacizumab Q2W Total group. | 2590 (1920) | NA (NA) — Cohort TT2A (participants with bevacizumab-refractory glioma), was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort TT2A (participants with bevacizumab-refractory glioma), was part of the MEDI3617 + Bevacizumab Q2W Total group.
  Cohort MP1 (n=7) | NA (NA) — Cohort MP1 was part of the MEDI3617 + Paclitaxel group. | NA (NA) — Cohort MP1 was part of the MEDI3617 + Paclitaxel group. | NA (NA) — Cohort MP1 was part of the MEDI3617 + Paclitaxel group. | 551 (331) | NA (NA) — Cohort MP1 was part of the MEDI3617 + Paclitaxel group.
  Cohort MP2 (n=6) | NA (NA) — Cohort MP2 was part of the MEDI3617 + Paclitaxel group. | NA (NA) — Cohort MP2 was part of the MEDI3617 + Paclitaxel group. | NA (NA) — Cohort MP2 was part of the MEDI3617 + Paclitaxel group. | 1460 (484) | NA (NA) — Cohort MP2 was part of the MEDI3617 + Paclitaxel group.
  Cohort MCP1 (n=4) | NA (NA) — Cohort MCP1 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP1 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP1 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP1 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | 1240 (882)
  Cohort MCP2 (n=3) | NA (NA) — Cohort MCP2 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP2 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP2 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP2 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | 2890 (257)

10. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) of MEDI3617
Description: The AUC0-inf is the Area Under the Concentration-Time Curve From Time Zero to infinity of MEDI3617. Here, "n" is number of participants analyzed for this endpoint at a specific dose.
Time Frame: as for outcome 8
Population: All participants who received treatment with MEDI3617 and for whom PK blood samples were collected and evaluated.
Measure: Mean (Standard Deviation); unit: day*mcg/mL
Arm/Group | MEDI3617 SINGLE AGENT TOTAL | MEDI3617 + BEVACIZUMAB Q3W ESCALATION TOTAL | MEDI3617 + BEVACIZUMAB Q2W TOTAL | MEDI3617 + PACLITAXEL TOTAL | MEDI3617 + CARBOPLATIN/PACLITAXEL TOTAL
Number analyzed (Participants) | 25 | 8 | 13 | 4 | 3
day*mcg/mL
  Cohort -2 (n=1) | 1.79 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort -2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort -2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort -2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort -2 was part of the MEDI3617 Single agent total group.
  Cohort 1 (n=1) | 8.12 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort 1 was part of the MEDI3617 Single agent total group | NA (NA) — Cohort 1 was part of the MEDI3617 Single agent total group | NA (NA) — Cohort 1 was part of the MEDI3617 Single agent total group | NA (NA) — Cohort 1 was part of the MEDI3617 Single agent total group
  Cohort 2 (n=2) | 269 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort 2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 2 was part of the MEDI3617 Single agent total group.
  Cohort 3 (n=3) | 529 (269) | NA (NA) — Cohort 3 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 3 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 3 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 3 was part of the MEDI3617 Single agent total group.
  Cohort 4 (n=2) | 2150 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort 4 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 4 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 4 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 4 was part of the MEDI3617 Single agent total group.
  Cohort 5 (n=2) | 4230 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort 5 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 5 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 5 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 5 was part of the MEDI3617 Single agent total group.
  Cohort OCE -1 (n=12) | 3280 (1410) | NA (NA) — Cohort OCE -1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE -1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE -1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE -1 was part of the MEDI3617 Single agent total group.
  Cohort OCE 1 (n=2) | 2490 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort OCE 1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE 1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE 1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE 1 was part of the MEDI3617 Single agent total group.
  Cohort MB 1A (n=3) | NA (NA) — Cohort MB 1A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | 110 (58.1) | NA (NA) — Cohort MB 1A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 1A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 1A was part of the MEDI3617 + Bevacizumab Q3W escalation group.
  Cohort MB 2A (n=3) | NA (NA) — Cohort MB 2A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | 628 (376) | NA (NA) — Cohort MB 2A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 2A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 2A was part of the MEDI3617 + Bevacizumab Q3W escalation group.
  Cohort MB 4A (n=2) | NA (NA) — Cohort MB 4A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | 3920 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort MB 4A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 4A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 4A was part of the MEDI3617 + Bevacizumab Q3W escalation group.
  Cohort MB 1B (n=7) | NA (NA) — Cohort MB 1B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 1B was part of the MEDI3617 + Bevacizumab Q2W Total group. | 104 (61) | NA (NA) — Cohort MB 1B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 1B was part of the MEDI3617 + Bevacizumab Q2W Total group.
  Cohort MB 2B (n=3) | NA (NA) — Cohort MB 2B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 2B was part of the MEDI3617 + Bevacizumab Q2W Total group. | 252 (83.2) | NA (NA) — Cohort MB 2B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 2B was part of the MEDI3617 + Bevacizumab Q2W Total group.
  Cohort MB 3B (n=2) | NA (NA) — Cohort MB 3B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 3B was part of the MEDI3617 + Bevacizumab Q2W Total group. | 1200 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort MB 3B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 3B was part of the MEDI3617 + Bevacizumab Q2W Total group.
  Cohort MB 4B (n=1) | NA (NA) — Cohort MB 4B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 4B was part of the MEDI3617 + Bevacizumab Q2W Total group. | 4630 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort MB 4B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 4B was part of the MEDI3617 + Bevacizumab Q2W Total group.
  Cohort MP1 (n=3) | NA (NA) — Cohort MP1 was part of the MEDI3617 + Paclitaxel group. | NA (NA) — Cohort MP1 was part of the MEDI3617 + Paclitaxel group. | NA (NA) — Cohort MP1 was part of the MEDI3617 + Paclitaxel group. | 849 (163) | NA (NA) — Cohort MP1 was part of the MEDI3617 + Paclitaxel group.
  Cohort MP2 (n=1) | NA (NA) — Cohort MP2 was part of the MEDI3617 + Paclitaxel group. | NA (NA) — Cohort MP2 was part of the MEDI3617 + Paclitaxel group. | NA (NA) — Cohort MP2 was part of the MEDI3617 + Paclitaxel group. | 2810 (NA) — Cohort MP2 was part of the MEDI3617 + Paclitaxel group. | NA (NA) — Cohort MP2 was part of the MEDI3617 + Paclitaxel group.
  Cohort MCP1 (n=1) | NA (NA) — Cohort MCP1 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP1 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP1 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP1 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | 2240 (NA) — Standard deviation was not calculated due to limited sample size (n<3).
  Cohort MCP2 (n=2) | NA (NA) — Cohort MCP2 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP2 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP2 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP2 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | 3560 (NA) — Standard deviation was not calculated due to limited sample size (n<3).

11. Secondary Outcome: Systemic Clearance (CL) of MEDI3617
Description: Systemic clearance describes the removal of drug from a volume of serum in a given unit of time (drug loss from the body). It is measured as milliliter per day (mL/day). Here, "n" is number of participants analyzed for this endpoint at a specific dose.
Time Frame: as for outcome 8
Population: All participants who received treatment with MEDI3617 and for whom PK blood samples were collected and evaluated.
Measure: Mean (Standard Deviation); unit: milliliter per day (mL/day)
Arm/Group | MEDI3617 SINGLE AGENT TOTAL | MEDI3617 + BEVACIZUMAB Q3W ESCALATION TOTAL | MEDI3617 + BEVACIZUMAB Q2W TOTAL | MEDI3617 + PACLITAXEL TOTAL | MEDI3617 + CARBOPLATIN/PACLITAXEL TOTAL
Number analyzed (Participants) | 25 | 8 | 13 | 4 | 3
milliliter per day (mL/day)
  Cohort -2 (n=1) | 2790 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort -2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort -2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort -2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort -2 was part of the MEDI3617 Single agent total group.
  Cohort 1 (n=1) | 2460 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort 1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 1 was part of the MEDI3617 Single agent total group.
  Cohort 2 (n=2) | 423 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort 2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 2 was part of the MEDI3617 Single agent total group.
  Cohort 3 (n=3) | 679 (345) | NA (NA) — Cohort 3 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 3 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 3 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 3 was part of the MEDI3617 Single agent total group.
  Cohort 4 (n=2) | 465 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort 4 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 4 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 4 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 4 was part of the MEDI3617 Single agent total group.
  Cohort 5 (n=2) | 355 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort 5 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 5 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 5 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 5 was part of the MEDI3617 Single agent total group.
  Cohort OCE -1 (n=12) | 352 (136) | NA (NA) — Cohort OCE -1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE -1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE -1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE -1 was part of the MEDI3617 Single agent total group.
  Cohort OCE 1 (n=2) | 603 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort OCE 1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE 1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE 1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE 1 was part of the MEDI3617 Single agent total group.
  Cohort MB 1A (n=3) | NA (NA) — Cohort MB 1A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | 1060 (426) | NA (NA) — Cohort MB 1A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 1A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 1A was part of the MEDI3617 + Bevacizumab Q3W escalation group.
  Cohort MB 2A (n=3) | NA (NA) — Cohort MB 2A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | 614 (363) | NA (NA) — Cohort MB 2A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 2A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 2A was part of the MEDI3617 + Bevacizumab Q3W escalation group.
  Cohort MB 4A (n=2) | NA (NA) — Cohort MB 4A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | 388 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort MB 4A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 4A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 4A was part of the MEDI3617 + Bevacizumab Q3W escalation group.
  Cohort MB 1B (n=7) | NA (NA) — Cohort MB 1B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 1B was part of the MEDI3617 + Bevacizumab Q2W Total group. | 797 (499) | NA (NA) — Cohort MB 1B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 1B was part of the MEDI3617 + Bevacizumab Q2W Total group.
  Cohort MB 2B (n=3) | NA (NA) — Cohort MB 2B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 2B was part of the MEDI3617 + Bevacizumab Q2W Total group. | 847 (237) | NA (NA) — Cohort MB 2B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 2B was part of the MEDI3617 + Bevacizumab Q2W Total group.
  Cohort MB 3B(n=2) | NA (NA) — Cohort MB 3B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 3B was part of the MEDI3617 + Bevacizumab Q2W Total group. | 501 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort MB 3B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 3B was part of the MEDI3617 + Bevacizumab Q2W Total group.
  Cohort MB 4B (n=1) | NA (NA) — Cohort MB 4B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 4B was part of the MEDI3617 + Bevacizumab Q2W Total group. | 216 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort MB 4B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 4B was part of the MEDI3617 + Bevacizumab Q2W Total group.
  Cohort MP1 (n=3) | NA (NA) — Cohort MP1 was part of the MEDI3617 + Paclitaxel group. | NA (NA) — Cohort MP1 was part of the MEDI3617 + Paclitaxel group. | NA (NA) — Cohort MP1 was part of the MEDI3617 + Paclitaxel group. | 727 (157) | NA (NA) — Cohort MP1 was part of the MEDI3617 + Paclitaxel group.
  Cohort MP2 (n=1) | NA (NA) — Cohort MP2 was part of the MEDI3617 + Paclitaxel group. | NA (NA) — Cohort MP2 was part of the MEDI3617 + Paclitaxel group. | NA (NA) — Cohort MP2 was part of the MEDI3617 + Paclitaxel group. | 356 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort MP2 was part of the MEDI3617 + Paclitaxel group.
  Cohort MCP1 (n=1) | NA (NA) — Cohort MCP1 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP1 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP1 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP1 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | 446 (NA) — Standard deviation was not calculated due to limited sample size (n<3).
  Cohort MCP2 (n=2) | NA (NA) — Cohort MCP2 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP2 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP2 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP2 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | 424 (NA) — Standard deviation was not calculated due to limited sample size (n<3).

12. Secondary Outcome: Terminal Elimination Half Life (t1/2) of MEDI3617
Description: The t1/2 is the time in days required for the concentration of the drug to reach half of its original value. Here, "n" is number of participants analyzed for this endpoint at a specific dose.
Time Frame: as for outcome 8
Population: All participants who received treatment with MEDI3617 and for whom PK blood samples were collected and evaluated.
Measure: Mean (Standard Deviation); unit: day
Arm/Group | MEDI3617 SINGLE AGENT TOTAL | MEDI3617 + BEVACIZUMAB Q3W ESCALATION TOTAL | MEDI3617 + BEVACIZUMAB Q2W TOTAL | MEDI3617 + PACLITAXEL TOTAL | MEDI3617 + CARBOPLATIN/PACLITAXEL TOTAL
Number analyzed (Participants) | 25 | 8 | 13 | 4 | 3
day
  Cohort -2 (n=1) | 0.585 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort -2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort -2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort -2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort -2 was part of the MEDI3617 Single agent total group.
  Cohort 1 (n=1) | 1.26 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort 1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 1 was part of the MEDI3617 Single agent total group.
  Cohort 2 (n=2) | 5.86 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort 2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 2 was part of the MEDI3617 Single agent total group.
  Cohort 3 (n=3) | 5.98 (3.09) | NA (NA) — Cohort 3 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 3 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 3 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 3 was part of the MEDI3617 Single agent total group.
  Cohort 4 (n=2) | 7.68 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort 4 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 4 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 4 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 4 was part of the MEDI3617 Single agent total group.
  Cohort 5 (n=2) | 7.79 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort 5 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 5 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 5 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 5 was part of the MEDI3617 Single agent total group.
  Cohort OCE -1 (n=12) | 10.4 (3.15) | NA (NA) — Cohort OCE -1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE -1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE -1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE -1 was part of the MEDI3617 Single agent total group.
  Cohort OCE 1 (n=2) | 9.03 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort OCE 1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE 1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE 1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE 1 was part of the MEDI3617 Single agent total group.
  Cohort MB 1A (n=3) | NA (NA) — Cohort MB 1A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | 3.59 (0.983) | NA (NA) — Cohort MB 1A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 1A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 1A was part of the MEDI3617 + Bevacizumab Q3W escalation group.
  Cohort MB 2A (n=3) | NA (NA) — Cohort MB 2A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | 9.67 (3.35) | NA (NA) — Cohort MB 2A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 2A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 2A was part of the MEDI3617 + Bevacizumab Q3W escalation group.
  Cohort MB 4A (n=2) | NA (NA) — Cohort MB 4A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | 12.3 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort MB 4A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 4A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 4A was part of the MEDI3617 + Bevacizumab Q3W escalation group.
  Cohort MB 1B (n=7) | NA (NA) — Cohort MB 1B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 1B was part of the MEDI3617 + Bevacizumab Q2W Total group. | 3.9 (2.69) | NA (NA) — Cohort MB 1B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 1B was part of the MEDI3617 + Bevacizumab Q2W Total group.
  Cohort MB 2B (n=3) | NA (NA) — Cohort MB 2B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 2B was part of the MEDI3617 + Bevacizumab Q2W Total group. | 5.12 (0.541) | NA (NA) — Cohort MB 2B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 2B was part of the MEDI3617 + Bevacizumab Q2W Total group.
  Cohort MB 3B(n=2) | NA (NA) — Cohort MB 3B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 3B was part of the MEDI3617 + Bevacizumab Q2W Total group. | 8.23 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort MB 3B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 3B was part of the MEDI3617 + Bevacizumab Q2W Total group.
  Cohort MB 4B (n=1) | NA (NA) — Cohort MB 4B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 4B was part of the MEDI3617 + Bevacizumab Q2W Total group. | 10.2 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort MB 4B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 4B was part of the MEDI3617 + Bevacizumab Q2W Total group.
  Cohort MP1 (n=3) | NA (NA) — Cohort MP1 was part of the MEDI3617 + Paclitaxel group. | NA (NA) — Cohort MP1 was part of the MEDI3617 + Paclitaxel group. | NA (NA) — Cohort MP1 was part of the MEDI3617 + Paclitaxel group. | 6.96 (1.59) | NA (NA) — Cohort MP1 was part of the MEDI3617 + Paclitaxel group.
  Cohort MP2 (n=1) | NA (NA) — Cohort MP2 was part of the MEDI3617 + Paclitaxel group. | NA (NA) — Cohort MP2 was part of the MEDI3617 + Paclitaxel group. | NA (NA) — Cohort MP2 was part of the MEDI3617 + Paclitaxel group. | 9.34 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort MP2 was part of the MEDI3617 + Paclitaxel group.
  Cohort MCP1 (n=1) | NA (NA) — Cohort MCP1 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP1 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP1 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP1 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | 15.1 (NA) — Standard deviation was not calculated due to limited sample size (n<3).
  Cohort MCP2 (n=2) | NA (NA) — Cohort MCP2 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP2 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP2 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP2 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | 11.1 (NA) — Standard deviation was not calculated due to limited sample size (n<3).

13. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibody (ADA)
Description: The immunogenic potential of MEDI3617 was assessed by summarizing the number and percentage of participants who develop detectable ADA. Immunogenicity assessment included determination of anti-drug (MEDI3617) antibodies in serum samples. Samples were measured for the presence of ADA using validated immunoassays.
Time Frame: Presence of ADA to MEDI3617 were assessed prior to infusion with MEDI3617 on Day 1 of each dosing cycle, as well as the end of treatment, and 30 days, 3 months, and 6 months post last dose of MEDI3617
Population: All participants who received treatment with MEDI3617.
Measure: Number; unit: participants
Arm/Group | MEDI3617 SINGLE AGENT TOTAL | MEDI3617 + BEVACIZUMAB Q3W ESCALATION TOTAL | MEDI3617 + BEVACIZUMAB Q2W TOTAL | MEDI3617 + PACLITAXEL TOTAL | MEDI3617 + CARBOPLATIN/PACLITAXEL TOTAL
Number analyzed (Participants) | 42 | 16 | 38 | 13 | 7
participants | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response rate defined as the number of participants with confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. CR was defined as disappearance of all target lesions, any pathological lymph nodes must have reduction in short axis to less than (<) 10 millimeter (the sum may not be "0" if there are target nodes). PR was defined as at least a 30 percent (%) decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Time from the first dose of investigational product until end of study
Population: Safety population included all participants who received treatment with MEDI3617.
Measure: Number; unit: Participants
Arm/Group | MEDI3617 SINGLE AGENT TOTAL | MEDI3617 + BEVACIZUMAB Q3W ESCALATION TOTAL | MEDI3617 + BEVACIZUMAB Q2W TOTAL | MEDI3617 + PACLITAXEL TOTAL | MEDI3617 + CARBOPLATIN/PACLITAXEL TOTAL
Number analyzed (Participants) | 42 | 16 | 38 | 13 | 7
Participants | 1 | 1 | 2 | 2 | 0

15. Secondary Outcome: Time to Response (TTR)
Description: Time to response (TTR) is defined as the time from the study entry to the first documentation of confirmed CR or confirmed PR. CR was defined as disappearance of all target lesions, any pathological lymph nodes must have reduction in short axis to less than (<) 10 millimeter (the sum may not be "0" if there are target nodes). PR was defined as at least a 30 percent (%) decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Analysis was based on responses confirmed at a repeat assessment made at least 4 weeks after the initial response, with the TTR taken as the first time the response was observed, not the confirmation assessment. TTR was evaluated using the Kaplan-Meier method.
Time Frame: Time from the first dose of investigational product until end of study
Population: Safety population included all participants who received treatment with MEDI3617.
Measure: Median (Full Range); unit: months
Arm/Group | MEDI3617 SINGLE AGENT TOTAL | MEDI3617 + BEVACIZUMAB Q3W ESCALATION TOTAL | MEDI3617 + BEVACIZUMAB Q2W TOTAL | MEDI3617 + PACLITAXEL TOTAL | MEDI3617 + CARBOPLATIN/PACLITAXEL TOTAL
Number analyzed (Participants) | 42 | 16 | 38 | 13 | 7
months | 2.6 [2.6 to 2.6] | 1.2 [1.2 to 1.2] | 2.0 [1.6 to 2.3] | 1.7 [1.6 to 1.7] | NA [NA to NA] — No objective response was observed in the MEDI3617 + carboplatin/paclitaxel cohorts.

16. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response is defined as the duration from the first documentation of objective disease response (ie, confirmed CR or confirmed PR) to the first documented disease progression. The duration of response was censored on the date of last tumor assessment documenting absence of disease progression for participants who have no documented progression prior to data cutoff, dropout, or the initiation of alternate anticancer treatment. Duration of response was evaluated for the subgroup of participants with an objective response using the Kaplan-Meier method.
Time Frame: Time from the first dose of investigational product until end of study
Population: Safety population included all participants who received treatment with MEDI3617.
Measure: Median (Full Range); unit: months
Arm/Group | MEDI3617 SINGLE AGENT TOTAL | MEDI3617 + BEVACIZUMAB Q3W ESCALATION TOTAL | MEDI3617 + BEVACIZUMAB Q2W TOTAL | MEDI3617 + PACLITAXEL TOTAL | MEDI3617 + CARBOPLATIN/PACLITAXEL TOTAL
Number analyzed (Participants) | 42 | 16 | 38 | 13 | 7
months | 3.7 [3.7 to 3.7] | NA [17.8 to 17.8] — Due to the lack of available data caused by censoring subjects in the MEDI3617 + bevacizumab Q3W escalation cohorts for this endpoint, median duration of response was not calculable. | NA [2.9 to 3.7] — Due to the lack of available data caused by censoring subjects in the MEDI3617 + bevacizumab Q2W cohorts for this endpoint, median duration of response was not calculable. | NA [1.6 to 17.7] — Due to the lack of available data caused by censoring subjects in the MEDI3617 + paclitaxel cohorts for this endpoint, median duration of response was not calculable. | NA [NA to NA] — No objective response was observed in the MEDI3617 + carboplatin/paclitaxel cohorts.

17. Secondary Outcome: Time to Progression (TTP)
Description: Time to progression (TTP) is defined as time from the start of treatment with MEDI3617 until the documentation of disease progression. The TTP was censored on the date of last tumor assessment documenting absence of tumor progression for participants who have no documented progression prior to data cutoff, dropout, or the initiation of alternate anticancer treatment. Participants having no tumor assessments after the start of treatment with MEDI3617 had TTP censored on the first date of treatment with MEDI3617. TTP was evaluated using the Kaplan-Meier method.
Time Frame: Time from the first dose of investigational product until end of study
Population: Safety population included all participants who received treatment with MEDI3617.
Measure: Median (Full Range); unit: months
Arm/Group | MEDI3617 SINGLE AGENT TOTAL | MEDI3617 + BEVACIZUMAB Q3W ESCALATION TOTAL | MEDI3617 + BEVACIZUMAB Q2W TOTAL | MEDI3617 + PACLITAXEL TOTAL | MEDI3617 + CARBOPLATIN/PACLITAXEL TOTAL
Number analyzed (Participants) | 42 | 16 | 38 | 13 | 7
months | 1.4 [0.0 to 8.6] | 11.4 [0.0 to 39.4] | 1.8 [0.0 to 5.3] | 3.5 [0.0 to 19.4] | NA [0.0 to 4.0] — Due to the lack of available data caused by censoring subjects in the MEDI3617 + carboplatin/paclitaxel cohorts for this endpoint, median time to progression was not calculable.

18. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was measured from the start of treatment with MEDI3617 until the documentation of disease progression or death due to any cause, whichever occurred first. PFS was censored on the date of last tumor assessment documenting absence of tumor progression for participants who have no documented progression and were still alive prior to data cutoff, dropout, or the initiation of alternate anticancer treatment. Participants having no tumor assessments after the start of treatment with MEDI3617 had PFS censored on the first date of treatment with MEDI3617. PFS was evaluated using the Kaplan-Meier method.
Time Frame: Time from the first dose of investigational product until end of study
Population: Safety population included all participants who received treatment with MEDI3617.
Measure: Median (Full Range); unit: months
Arm/Group | MEDI3617 SINGLE AGENT TOTAL | MEDI3617 + BEVACIZUMAB Q3W ESCALATION TOTAL | MEDI3617 + BEVACIZUMAB Q2W TOTAL | MEDI3617 + PACLITAXEL TOTAL | MEDI3617 + CARBOPLATIN/PACLITAXEL TOTAL
Number analyzed (Participants) | 42 | 16 | 38 | 13 | 7
months | 1.4 [0.0 to 8.6] | 11.4 [0.0 to 39.4] | 1.7 [0.0 to 5.3] | 3.5 [0.0 to 19.4] | NA [0.0 to 4.0] — Due to the lack of available data caused by censoring subjects in the MEDI3617 + carboplatin/paclitaxel cohorts for this endpoint, median progression-free survival was not calculable.

19. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from the start of treatment with MEDI3617 until death. For the participants who were alive at the end of study or lost to follow-up, overall survival was censored on the last date when participants were known to be alive. Overall survival was evaluated using the Kaplan-Meier method.
Time Frame: Time from the first dose of investigational product until death due to any cause
Population: Safety population included all participants who received treatment with MEDI3617.
Measure: Median (Full Range); unit: months
Arm/Group | MEDI3617 SINGLE AGENT TOTAL | MEDI3617 + BEVACIZUMAB Q3W ESCALATION TOTAL | MEDI3617 + BEVACIZUMAB Q2W TOTAL | MEDI3617 + PACLITAXEL TOTAL | MEDI3617 + CARBOPLATIN/PACLITAXEL TOTAL
Number analyzed (Participants) | 42 | 16 | 38 | 13 | 7
months | 11.4 [0.3 to 46.8] | 25.7 [1.3 to 42.8] | 7.4 [0.5 to 33.4] | 14.2 [1.0 to 35.7] | NA [1.9 to 34.4] — Due to the lack of available data caused by censoring subjects in the MEDI3617 + carboplatin/paclitaxel cohorts for this endpoint, median overall survival was not calculable.

20. Secondary Outcome: Circulating Levels of Angiopoietin 2 (Ang2)
Description: Profile of Ang2 post MEDI3617 administration in relation to time course of antibody concentrations.
Time Frame: Prior to infusion on Cycle 4 and Cycle 5
Population: All participants who received treatment with MEDI3617 and for whom PD blood samples were collected and evaluated.
Measure: Mean (Standard Deviation); unit: nanogram per millileter (ng/mL)
Arm/Group | MEDI3617 SINGLE AGENT TOTAL | MEDI3617 + BEVACIZUMAB Q3W ESCALATION TOTAL | MEDI3617 + BEVACIZUMAB Q2W TOTAL | MEDI3617 + PACLITAXEL TOTAL | MEDI3617 + CARBOPLATIN/PACLITAXEL TOTAL
Number analyzed (Participants) | 14 | 11 | 7 | 3 | 2
nanogram per millileter (ng/mL)
  Cycle 4: Cohort -2 (n=2) | 4.07 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort -2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort -2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort -2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort -2 was part of the MEDI3617 Single agent total group.
  Cycle 5: Cohort -2 (n=2) | 4.28 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort -2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort -2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort -2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort -2 was part of the MEDI3617 Single agent total group.
  Cycle 4: Cohort -1 (n=2) | 5.11 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort -1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort -1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort -1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort -1 was part of the MEDI3617 Single agent total group.
  Cycle 4: Cohort 1 (n=3) | 5.69 (4.02) | NA (NA) — Cohort 1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 1 was part of the MEDI3617 Single agent total group.
  Cycle 5: Cohort 1 (n=2) | 8.22 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort 1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 1 was part of the MEDI3617 Single agent total group.
  Cycle 4: Cohort 2 (n=1) | 307.53 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort 2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 2 was part of the MEDI3617 Single agent total group.
  Cycle 5: Cohort 2 (n=1) | 924.66 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort 2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 2 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 2 was part of the MEDI3617 Single agent total group.
  Cycle 4: Cohort 3 (n=1) | 341.21 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort 3 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 3 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 3 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 3 was part of the MEDI3617 Single agent total group.
  Cycle 5: Cohort 3 (n=1) | 265.86 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort 3 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 3 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 3 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 3 was part of the MEDI3617 Single agent total group.
  Cycle 4: Cohort 4 (n=1) | 288.10 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort 4 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 4 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 4 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 4 was part of the MEDI3617 Single agent total group.
  Cycle 4: Cohort 5 (n=1) | 1181.14 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort 5 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 5 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 5 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 5 was part of the MEDI3617 Single agent total group.
  Cycle 5: Cohort 5 (n=1) | 1451.43 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort 5 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 5 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 5 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort 5 was part of the MEDI3617 Single agent total group.
  Cycle 4: Cohort OCE -1 (n=3) | 312.27 (151.19) | NA (NA) — Cohort OCE -1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE -1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE -1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE -1 was part of the MEDI3617 Single agent total group.
  Cycle 5: Cohort OCE -1 (n=3) | 206.43 (83.74) | NA (NA) — Cohort OCE -1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE -1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE -1 was part of the MEDI3617 Single agent total group. | NA (NA) — Cohort OCE -1 was part of the MEDI3617 Single agent total group.
  Cycle 4: Cohort MB 1A (n=2) | NA (NA) — Cohort MB 1A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | 386.13 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort MB 1A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 1A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 1A was part of the MEDI3617 + Bevacizumab Q3W escalation group.
  Cycle 5: Cohort MB 1A (n=2) | NA (NA) — Cohort MB 1A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | 421.74 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort MB 1A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 1A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 1A was part of the MEDI3617 + Bevacizumab Q3W escalation group.
  Cycle 4: Cohort MB 2A (n=3) | NA (NA) — Cohort MB 2A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | 215.71 (143.16) | NA (NA) — Cohort MB 2A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 2A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 2A was part of the MEDI3617 + Bevacizumab Q3W escalation group.
  Cycle 5: Cohort MB 2A (n=2) | NA (NA) — Cohort MB 2A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | 228.92 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort MB 2A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 2A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 2A was part of the MEDI3617 + Bevacizumab Q3W escalation group.
  Cycle 4: Cohort MB 3A (n=1) | NA (NA) — Cohort MB 3A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | 218.48 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort MB 3A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 3A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 3A was part of the MEDI3617 + Bevacizumab Q3W escalation group.
  Cycle 5: Cohort MB 3A (n=2) | NA (NA) — Cohort MB 3A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | 247.51 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort MB 3A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 3A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 3A was part of the MEDI3617 + Bevacizumab Q3W escalation group.
  Cycle 4: Cohort MB 4A (n=4) | NA (NA) — Cohort MB 4A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | 368.08 (257.59) | NA (NA) — Cohort MB 4A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 4A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 4A was part of the MEDI3617 + Bevacizumab Q3W escalation group.
  Cycle 5: Cohort MB 4A (n=2) | NA (NA) — Cohort MB 4A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | 353.73 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort MB 4A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 4A was part of the MEDI3617 + Bevacizumab Q3W escalation group. | NA (NA) — Cohort MB 4A was part of the MEDI3617 + Bevacizumab Q3W escalation group.
  Cycle 4: Cohort MB 1B (n=2) | NA (NA) — Cohort MB 1B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 1B was part of the MEDI3617 + Bevacizumab Q2W Total group. | 466.27 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort MB 1B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 1B was part of the MEDI3617 + Bevacizumab Q2W Total group.
  Cycle 5: Cohort MB 1B (n=1) | NA (NA) — Cohort MB 1B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 1B was part of the MEDI3617 + Bevacizumab Q2W Total group. | 750.61 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort MB 1B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 1B was part of the MEDI3617 + Bevacizumab Q2W Total group.
  Cycle 4: Cohort MB 2B (n=1) | NA (NA) — Cohort MB 2B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 2B was part of the MEDI3617 + Bevacizumab Q2W Total group. | 421.03 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort MB 2B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 2B was part of the MEDI3617 + Bevacizumab Q2W Total group.
  Cycle 5: Cohort MB 2B (n=1) | NA (NA) — Cohort MB 2B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 2B was part of the MEDI3617 + Bevacizumab Q2W Total group. | 387.45 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort MB 2B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 2B was part of the MEDI3617 + Bevacizumab Q2W Total group.
  Cycle 4:Cohort MB 3B (n=1) | NA (NA) — Cohort MB 3B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 3B was part of the MEDI3617 + Bevacizumab Q2W Total group. | 141.93 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort MB 3B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 3B was part of the MEDI3617 + Bevacizumab Q2W Total group.
  Cycle 4: Cohort MB 4B (n=3) | NA (NA) — Cohort MB 4B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 4B was part of the MEDI3617 + Bevacizumab Q2W Total group. | 229.19 (109.02) | NA (NA) — Cohort MB 4B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 4B was part of the MEDI3617 + Bevacizumab Q2W Total group.
  Cycle 5: Cohort MB 4B (n=1) | NA (NA) — Cohort MB 4B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 4B was part of the MEDI3617 + Bevacizumab Q2W Total group. | 174.65 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort MB 4B was part of the MEDI3617 + Bevacizumab Q2W Total group. | NA (NA) — Cohort MB 4B was part of the MEDI3617 + Bevacizumab Q2W Total group.
  Cycle 4: Cohort MP1 (n=1) | NA (NA) — Cohort MP1 was part of the MEDI3617 + Paclitaxel group. | NA (NA) — Cohort MP1 was part of the MEDI3617 + Paclitaxel group. | NA (NA) — Cohort MP1 was part of the MEDI3617 + Paclitaxel group. | 339.35 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort MP1 was part of the MEDI3617 + Paclitaxel group.
  Cycle 4: Cohort MP2 (n=2) | NA (NA) — Cohort MP2 was part of the MEDI3617 + Paclitaxel group. | NA (NA) — Cohort MP2 was part of the MEDI3617 + Paclitaxel group. | NA (NA) — Cohort MP2 was part of the MEDI3617 + Paclitaxel group. | 210.43 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort MP2 was part of the MEDI3617 + Paclitaxel group.
  Cycle 5: Cohort MP2 (n=2) | NA (NA) — Cohort MP2 was part of the MEDI3617 + Paclitaxel group. | NA (NA) — Cohort MP2 was part of the MEDI3617 + Paclitaxel group. | NA (NA) — Cohort MP2 was part of the MEDI3617 + Paclitaxel group. | 166.73 (NA) — Standard deviation was not calculated due to limited sample size (n<3). | NA (NA) — Cohort MP2 was part of the MEDI3617 + Paclitaxel group.
  Cycle 4: Cohort MCP1 (n=2) | NA (NA) — Cohort MCP1 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP1 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP1 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP1 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | 348.53 (NA) — Standard deviation was not calculated due to limited sample size (n<3).
  Cycle 5: Cohort MCP1 (n=2) | NA (NA) — Cohort MCP1 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP1 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP1 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | NA (NA) — Cohort MCP1 was part of the MEDI3617 + Carboplatin/Paclitaxel group. | 336.31 (NA) — Standard deviation was not calculated due to limited sample size (n<3).

21. Primary Outcome: Number of Participants With a Decline in Karnofsky Performance Status (KPS) of ≥ 20 Points at Worst Record On-study Compared With Baseline
Description: KPS scale: 100 is no evidence of disease; 90 is able to carry on normal activity, minor symptoms of disease; 80 is normal activity with effort, some symptoms of disease; 70 is cares for self; unable to do active work; 60 is requires occasional assistance, but is able to care for most of his needs; 50 is requires considerable assistance with frequent medical care; 40 is disabled, requires special care; 30 is severely disabled, hospitalization is indicated although death is not imminent; 20 is very sick, hospitalization necessary, active support treatment necessary; 10 is moribund, fatal processes progressing rapidly, 0 is dead.
Time Frame: From start of study drug administration up to 30 days after the last dose of MEDI3617
Population: Safety population included all participants who received treatment with MEDI3617
Measure: Number; unit: Participants
Arm/Group | MEDI3617 SINGLE AGENT TOTAL | MEDI3617 + BEVACIZUMAB Q3W ESCALATION TOTAL | MEDI3617 + BEVACIZUMAB Q2W TOTAL | MEDI3617 + PACLITAXEL TOTAL | MEDI3617 + CARBOPLATIN/PACLITAXEL TOTAL
Number analyzed (Participants) | 42 | 16 | 38 | 13 | 7
Participants | 11 | 6 | 7 | 1 | 1

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to 90 days after the last dose of MEDI3617
Arm/Group | MEDI3617 SINGLE AGENT TOTAL | MEDI3617 + BEVACIZUMAB Q3W ESCALATION TOTAL | MEDI3617 + BEVACIZUMAB Q2W TOTAL | MEDI3617 + PACLITAXEL TOTAL | MEDI3617 + CARBOPLATIN/PACLITAXEL TOTAL
Serious Adverse Events (participants affected / at risk) | 18/42 | 4/16 | 18/38 | 7/13 | 4/7
Other Adverse Events (participants affected / at risk) | 40/42 | 16/16 | 34/38 | 13/13 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI3617 SINGLE AGENT TOTAL (N=42) | MEDI3617 + BEVACIZUMAB Q3W ESCALATION TOTAL (N=16) | MEDI3617 + BEVACIZUMAB Q2W TOTAL (N=38) | MEDI3617 + PACLITAXEL TOTAL (N=13) | MEDI3617 + CARBOPLATIN/PACLITAXEL TOTAL (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Faecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical device pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI3617 SINGLE AGENT TOTAL (N=42) | MEDI3617 + BEVACIZUMAB Q3W ESCALATION TOTAL (N=16) | MEDI3617 + BEVACIZUMAB Q2W TOTAL (N=38) | MEDI3617 + PACLITAXEL TOTAL (N=13) | MEDI3617 + CARBOPLATIN/PACLITAXEL TOTAL (N=7)
Anaemia (Blood and lymphatic system disorders) | 4 (5) | 1 (1) | 1 (1) | 2 (2) | 2 (3)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vision blurred (Eye disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 2 (2) | 3 (3) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 16 (19) | 9 (12) | 4 (4) | 4 (6) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 8 (11) | 5 (7) | 3 (4) | 4 (4) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 7 (7) | 2 (3) | 1 (1) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 11 (13) | 8 (14) | 11 (13) | 4 (6) | 4 (5)
Vomiting (Gastrointestinal disorders) | 11 (14) | 5 (8) | 3 (5) | 2 (2) | 2 (3)
Chills (General disorders) | 4 (4) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Fatigue (General disorders) | 18 (26) | 10 (13) | 12 (13) | 5 (6) | 3 (5)
Mucosal inflammation (General disorders) | 2 (2) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 11 (15) | 2 (12) | 7 (16) | 4 (7) | 0 (0)
Pyrexia (General disorders) | 2 (3) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Weight increased (Investigations) | 8 (11) | 2 (15) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 8 (11) | 5 (6) | 5 (7) | 1 (3) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (6) | 2 (2) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (8) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 4 (4) | 1 (2) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 4 (9) | 2 (2) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 8 (10) | 4 (4) | 1 (2) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 13 (14) | 7 (10) | 2 (2) | 2 (6) | 1 (1)
Dysgeusia (Nervous system disorders) | 4 (5) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 7 (8) | 4 (6) | 7 (8) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 4 (4) | 2 (2) | 3 (5) | 4 (5) | 2 (2)
Paraesthesia (Nervous system disorders) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3) | 4 (6) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 4 (5) | 4 (4) | 2 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (5) | 1 (3) | 5 (14) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 4 (5) | 2 (3) | 2 (2) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 3 (4) | 4 (4) | 3 (3) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (5) | 2 (3) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (4) | 0 (0) | 3 (4) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 10 (12) | 6 (24) | 13 (16) | 3 (3) | 2 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
"MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome" in the agreement description.